CLINICAL TRIAL: NCT06191705
Title: Urdu Translation, Validity and Reliability of Quick Disabilities of Arm, Shoulder & Hand (QuickDASH)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Other Study IDs: FUI/CTR/2023/26
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Arm, Shoulder or Hand pain /symptoms.
  Interventions: Diagnostic Test: QuickDASH

INTERVENTIONS:
Diagnostic Test: QuickDASH — Participants will be administered Urdu version of QuickDASH to collect data regarding Disabilities of Arm, Shoulder & Hand twice with a time interval of 72 hours to determine validity and reliability.

SUMMARY:
The purpose of this study is to translate Quick Disabilities of Arm, Shoulder & Hand (QuickDASH) into Urdu and determine the validity and reliability of the Urdu version of QuickDASH.

ELIGIBILITY:
Inclusion Criteria:

Individuals with for shoulder, arm/wrist, or hand musculoskeletal injury/pain/symptoms. Capable of understanding and completing the self-reported questionnaires. The exclusion criteria were the -

Exclusion Criteria:

Presence of any systemic disease or any neurological disorder. The upper limb involvement is due to any recent surgery in less than 6 weeks.

-

Ages: 19 Years to 44 Years | Sex: All
Age Groups: Adult
Study Population: Individuals with for shoulder, arm/wrist, or hand musculoskeletal injury/pain/symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
QuickDASH | 72 hours
  Quick Disabilities of Arm, Shoulder & Hand (QuickDASH) is used to determine the Disabilities of Arm, Shoulder and Hand. A higher score signifies poor outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No